CLINICAL TRIAL: NCT04453072
Title: Behavioral Weight Loss Intervention Utilizing Mobile Health Technology in Hematopoietic Stem Cell Transplant Patients (BWL001)
Brief Title: A Study to See if an iPhone Weight Management App Can Help Promote Weight Loss in Adolescents and Young Adults After a Stem Cell Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: eHealth International, INC. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-001992; NCI-2020-02687 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-06-10; First posted 2020-07-01 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Malignant Neoplasm
MeSH Terms: conditions — Obesity; Neoplasms | interventions — Interviews as Topic; Weights and Measures; Spermine Synthase; Communication Devices for People with Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (app, scales, coaching, questionnaire) (Experimental): Patients receive an iPhone with W8Loss2Go app, a body scale and a digital food scale to weigh themselves and food daily. Patients interact with coaches via text messages for 4 days weekly and receive weekly 15 minute phone calls for appointment reminders, emotional support, progress discussion, and follow up on items discussed in a prior visit or phone call. Patients also have telemedicine interviews with the coach lasting 60 minutes at 2 and 4 months to elicit both positive and negative impacts on weight management and to identify barriers such as emotional eating, displacement behaviors, poor coping skills to life stressors, and social challenges. Patients who opt to extend the intervention until month 12 attend an additional telemedicine meeting with the coach. Patients also complete questionnaires over approximately 1.5 hours.
  Interventions: Other: Interview; Other: Media Intervention; Other: Questionnaire Administration; Other: Scale Device; Behavioral: Telephone-Based Intervention; Other: Text Message

INTERVENTIONS:
Other: Interview — Participate in interviews
Other: Media Intervention — Receive iPhone with W8Loss2Go app
Other: Questionnaire Administration — Complete questionnaires
Other: Scale Device — Receive body scale and food scale
  Other Names: Scale
Behavioral: Telephone-Based Intervention — Receive telephone calls
Other: Text Message — Receive text message
  Other Names: Short Message Service (SMS) Text; SMS Text Message; Text

SUMMARY:
This early phase I trial studies how well a behavioral weight loss intervention consisting of a smartphone application and coaching works for the promotion of weight loss in adolescents and young adults after a stem cell transplant. This study may help researchers learn more about how adolescents and young adults can lose weight and develop healthy eating habits.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effectiveness of an addiction-based weight loss intervention, embodied as a smartphone application (app) with telephone coaching, on weight outcomes of overweight and obese post hematopoietic stem cell transplantation (HSCT) adolescents and young adults.

SECONDARY OBJECTIVES:

I. To evaluate the changes in metabolic parameters and physical activity levels, in addition to modifications in addictive eating behaviors, motivation, and self-regulatory behaviors.

II. To evaluate the feasibility, adherence, and satisfaction of this intervention.

OUTLINE:

Patients receive an iPhone with W8Loss2Go app, a body scale and a digital food scale to weigh themselves and food daily. Patients interact with coaches via text messages for 4 days weekly and receive weekly 15 minute phone calls for appointment reminders, emotional support, progress discussion, and follow up on items discussed in a prior visit or phone call. Patients also have telemedicine interviews with the coach lasting 60 minutes at 2 and 4 months to elicit both positive and negative impacts on weight management and to identify barriers such as emotional eating, displacement behaviors, poor coping skills to life stressors, and social challenges. Patients who opt to extend the intervention until month 12 attend an additional telemedicine meeting with the coach. Patients also complete questionnaires over approximately 1.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of HSCT of any type, at least 100 days post-transplant at initial consultation of the study, will be eligible for the study
* Patients must classify as obese, represented as body mass index (BMI) >= 85th percentile for age and gender
* Patients must also be able to read English since the app intervention is only available in English form
* No patients will be excluded for any specific underlying medical condition, but decisions will be made on a case by case basis if a patient's functioning is deemed to significantly interfere with intervention participation
* PARENT:
* His/her child meets all inclusion criteria
* >= 18 years of age
* Can speak English

Exclusion Criteria:

* Patients who are < 100 days post-transplant at initial consultation will not be eligible for the study, but may become eligible if they are > 100 days post-transplant at their next consultation that falls within the enrollment window
* Patients whose BMI does not fall under the obese category will be excluded

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index (BMI) status | Baseline up to 12 months
  The main outcomes measures will be height (meters), weight (kg), and BMI (kg/m^2). Height will be measured to assess consistency in height measurements. Weight will be measured to assess trends in weight over the time span of the intervention. BMI will be measured as a product of weight and height to obtain an appropriate metric that accounts for these measures, and is the standard measure to assess weight progression in weight intervention studies.

SECONDARY OUTCOMES:
Adherence | Up to 12 months
  Compliance with app intervention will be measured by daily interaction with the application and the coach. A point system has been designed in the application to measure compliance with the app intervention, measured by +/- weight measured daily, logging of problem foods, logging of snacking panel, and logging of meals. The coach interacts with the participants through text daily, and through phone calls weekly.
Fasting lab test analysis: HbA1c | At four months up to 12 months
  HbA1c: Glycated hemoglobin (A1C) test result reflects your average blood sugar level for the past two to three months. Specifically, the A1C test measures what percentage of your hemoglobin is coated with sugar. The healthy range is between 4% and 5.6%
Fasting lab test analysis: Total cholesterol | At four months up to 12 months
  Total cholesterol: This measures the overall amount of cholesterol in your blood. The healthy range is < 170 mg/dL
Fasting lab test analysis: Low density lipoprotein | At four months up to 12 months
  LDL: low density lipoprotein (LDL) is the bad cholesterol in your blood. The healthy range is <100 mg/dL
Fasting lab test analysis: High density lipoprotein | At four months up to 12 months
  HDL: high density lipoprotein (HDL) is the good cholesterol in your blood. The healthy range is > 45 mg/dL
Fasting lab test analysis: triglycerides | At four months up to 12 months
  TG: triglycerides (TG) are a type of lipid in your blood. The healthy range is < 150 mg/dL
Fasting lab test analysis: aspartate/alanine aminotransferase | At four months up to 12 months
  AST/ALT: aspartate/alanine aminotransferase (AST/ALT) are liver enzymes to measure liver health. The healthy range or AST is 10-34 IU/L and the healthy range for ALT is 8-37 IU/L.
Fasting lab test analysis: glucose | At four months up to 12 months
  Glucose: This measures the amount of sugar in your blood. We measure this after fasting for 8 hours. The healthy range is 70-99 mg/dL
Yale Food Addiction Scale | Up to 12 months
  visual analog scale (1: never to 5:always). Higher scores may suggest more addictive like eating
Center for epidemiologic studies depression scale | Up to 12 months
  4 categorical options (never/rarely, sometimes, moderately, all of the time). A higher score suggests utility for screening for depression
Perceived stress scale | Up to 12 months
  Likert Scale (0: never to 4:very often). Higher scores suggests higher stress
Satisfaction with program | Up to 12 months
  Measured by "Satisfaction Survey". This Likert Scale will be completed by the participant and their parent at the end of the study. This scale uses a Likert Scale where 1 = completely disagree to 7 = completely agree. Higher scores suggest greater satisfaction with the intervention.
Demographic questionnaire | Up to 12 months
  10 questions with varying options to inquire about common demographic questions (gender, age, primary language, etc). Questions are descriptive in nature and no score is assigned.
Food craving questionnaire | Up to 12 months
  Likert scale (1: never to 5: always). A higher score suggests higher degrees of food cravings
Binge eating disorder screen | Up to 12 months
  4 categorical options (never/rarely, sometimes, often, always). A higher score suggests utility for screening for binge eating disorder
Physical activity questionnaire | Up to 12 months
  participants identify number of times (0 to more than 7) that they conducted a particular physical activity in the past 7 days. This includes skipping, rowing, etc.
S weight | Up to 12 months
  Likert scale (1: strongly disagree to 5: strongly agree). Higher scores indicates more motivation for change in weight
Height encounters questionnaire | Up to 12 months
  six questions about the participants health care utilization in the past month. Questions are descriptive in nature and no score is assigned.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore B Moore, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States